Previvors Recharge: A Resilience Program for Cancer Previvors (PreCharge)

NCT06378749

Statistical Analysis Plan: R43CA275673

March 21, 2023

## Statistical Analysis Plan

This study involved a single-group, pre-post design. Paired t-tests were used to determine the effect of the *PreCharge* intervention on the primary and secondary outcomes. The primary outcome was change, from pretest (baseline) to posttest (30 day follow-up), in resilience as measured by the Connor Davidson Resilience Scale (CDRISC-10). Secondary outcome measures include change in psychological flexibility (as measured by the Acceptance and Action Questionnaire – version 2 (AAQII). between pretest (baseline) and posttest (30 day follow-up) assessments. Cohen's d was used to assess the magnitude of the differences.